CLINICAL TRIAL: NCT04425109
Title: Department of Nutrition Science, Medical Faculty, Universitas Diponegoro Semarang, Indonesia
Brief Title: The Effect of Fermented and Non-fermented Soy Based Food in Appetite and Satiety Biomarker Among Young Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Etika Ratna Noer, Department of Nutrition, Medical Faculty, Universitas Diponegoro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SOY
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Obesity, Abdominal; Weight Loss
Keywords: tempeh; appetite; satiety; obesity
MeSH Terms: conditions — Obesity, Abdominal; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: Group 1 : give tempeh steak Group 2 : give soybean steak washout 3 days Group 1 : give soybean steak Group 2 : give tempeh steak
Who Masked: Participant, Investigator
Masking Description: subject with random allocation Investigator do not know the group the analysator do not know the group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tempeh steak (Experimental): The subjects were received the tempeh steak meal with isocal diet containing energy 307.4Kcal
  Interventions: Behavioral: meal test response
- soybean steak (Experimental): The subjects were received the soybean steak meal with isocal diet containing energy 307.4Kcal
  Interventions: Behavioral: meal test response

INTERVENTIONS:
Behavioral: meal test response — soy fermented versus non fermented meal test

SUMMARY:
Limited data are available regarding the satiety effects from fermented and non-fermented soy-based food. The aim of this study was to compare fermented (tempeh) and non-fermented soy-based diets high in protein in increasing satiety. Thirteen young obese females were studied in single-blind and cross over design. Blood samples were assessed frequently for 0, 30 and 120 minutes after consumption of two isocaloric breakfast which consist of tempeh and non-fermented soybean content. The energy content was 27% protein, 21% fat and 52% carbohydrate. Subjective satiety score was recorded at 30 and 120 minutes after taking a meal. Compared to non-fermented soybean, tempeh showed a steady trend in postprandial ghrelin, significantly increasing insulin and arginine, and decreasing glucose at 120 minutes. Satiety scores had the same trend in the hunger and fullness aspects between the meals.

DETAILED DESCRIPTION:
1. Introduction Obesity is a complex metabolic condition thought to result from an imbalance in energy intake and energy expenditure that results in excess fat accumulation in various adipose tissues and organs. It has been proposed that managing the dietary composition may be an efficient way to reduce body weight.

   Ghrelin is a circulating orexigenic hormone involved in both short-term food intake control at single meal. Protein has the most suppressive effect as opposed to other macronutrients on food intake. It has also been shown that dietary protein induces greater satiation and weight loss than carbohydrates. Postprandial ghrelin and insulin responses have been shown to be lower in high dietary protein Soybeans provide one of the most plentiful dietary protein sources for plants varies from 36% to 56%. Soy protein is a complete protein since it contains most of the important amino acids found in animal proteins.

   Limited evidence from soybean related satiety study suggests that tempeh may have an important role in obesity prevention and weight loss through satiating effects when replacing other protein foods in a mixed diet.

   Thus far, there have been only limited data regarding the satiety effects of dietary soy protein vs fermented soy protein on obesity in humans. The study aimed to examine the effect of anorexigenic hormone response and subjective satiety underfermented and isocaloric soy-based protein diet
2. Methods and Matherials

2.1. Subjects The subjects were recruited from advertisement who were motivated enough to respond actively to the request for topics. We used the following exclusion criteria: 1) a clinically significant history of chronic diseases, such as cardiovascular disease, diabetes, dyslipidemia or hypertension; 2) use of a weight-related medication/food; 3) heavy alcohol/drug consumption; and 4) pregnancy, breastfeeding, or intention to become pregnant during the time of the study. The subjects were divided into the TD, which were given tempeh, and SD, which were given soy, groups, to receive the meal than a crossover. All subjects signed a written consent form before participating in the studies, which were approved by Kariadi Hospital-Medical Faculty of Diponegoro University.

2.2. Preparation of Meal Diets The ingredient contents of the tempeh steak and soybean steak are listed. Tempeh Steak including : Tempeh 100g, 50g potato, 50g carrot and 50g green peas. Soybean Steak : Soybean 100g, 50g potato, 50g carrot, 50g green peas. The energy content of both are 307.4 Calorie (21.7g Protein, 8g Fat, 42.3g Carbohydrate, 4.5g fiber)

2.3. Anthropometric measurement Body weight, height, and body fat mass, lean mass, andfat-freemass were collected by a bioelectric impedance analyzer (SECA). BMI was calculated as body weight in kilograms divided by height in meters squared (kg/m2). Waist Circumference (WC) was measured with ainelastic measuring tape aroundthe mid-section between the margin of the last rib and the iliac crest.

2.4. Biochemical analysis Blood samples were collected from subjects'forearms. Venous blood specimens were collected in EDTA-treated and plain tubes after a 12-h fast. Blood samples were collected at 0 (fasting), 60, and 180mins. One tube containing EDTA was collected for acyl ghrelin analyses and plain tube collected for arginine, glucose, and insulin analyses. The tubes were centrifuged at 3000 × g for 10 minutesat 4°C, separated into plasma or serum, and stored at -80°C untilanalysis. Serum concentrations of acyl ghrelin, insulin and arginine were measured using an enzyme-linked immunosorbent assay (ELISA)

2.5. Scoring of subjective satiety usingvisual analogue scales (VAS) Visual Analogue Scales Food intake motivation was assessed with 100 mm line. Participants completed VAS to measure hunger/fullness at the same time points that blood samples were taken throughout the study protocol (ie. 0, 30, 180 minutes). The VAS questionnaire provides a subjective assessment of appetite-related sensations over time and allows the relationship between biochemical and dietary intake data to be explored. Visual analogue scales have been found to be a reliable and valid method to assess subjective states related to food intake behavior. On each of the test days, participants were asked to rate the following components relating to hunger and satiety using various questions, scored using the VAS instrument: (1) Hunger: how hungry do you feel at this moment? (VAS1) (2) The desire to eat: how strong is your desire to eat at this moment? (VAS5- VAS8); (3) Fullness: how full does your stomach feel at this moment? (VAS2, VAS3); (4) Motivation to eat: how much food do you think you could eat at this moment? (VAS4)

2.6 Statistical Analysis Data were analyzed IBM SPSS. Variable not normally distributed were nonparametric test. Wann whitney U test was used to test for difference all parameter at baseline. We compared change in variable (baseline, 30, 180 minutes) in each sub group using pair t=test or wilcoxon signed rank test to determine the impact of differential change. To test for change in parameters between two group used kruskal wallis.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m2
* female

Exclusion Criteria:

* clinically significant history of chronic diseases, such as cardiovascular disease, diabetes, dyslipidemia or hypertension
* use of a weight-related medication/food;
* heavy alcohol/drug consumption;
* pregnancy and breastfeeding

Ages: 19 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
change acylated ghrelin | 1 days
  Change acyl ghrelin at 0, 30, and 180 minutes from venous blood, taken after meal intake
change glucose | 1 days
  Change glucose at 0, 30, and 180 minutes from venous blood, taken after meal intake
change arginine | 1 days
  Change arginine at 0, 30, and 180 minutes from venous blood, taken after meal intake
change insulin | 1 days
  Change insulin at 0, 30, and 180 minutes from venous blood, taken after meal intake
Visual Analogue scale (VAS) | 1 days
  VAS measure hunger/fullness at the same time points that blood samples were taken throughout the study protocol (ie. 0, 30, 180 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Etika Noer, Principal Investigator — Universitas Diponegoro
Locations (1):
- Etika Ratna Noer, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
the result of this study is available to cite everyone
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: etikaratna@fk.undip.ac.id
URL: http://dept-gizi@fk.undip.ac.id

REFERENCES:
- [Derived] Noer ER, Dewi L, Kuo CH. Fermented soybean enhances post-meal response in appetite-regulating hormones among Indonesian girls with obesity. Obes Res Clin Pract. 2021 Jul-Aug;15(4):339-344. doi: 10.1016/j.orcp.2021.06.005. Epub 2021 Jun 17. PMID 34147377